CLINICAL TRIAL: NCT06057558
Title: Studying the Airway Microbiome of Cystic Fibrosis Patients and the Potential of Probiotics for the Airways
Brief Title: Airway Microbiome of Cystic Fibrosis Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Kim Van Hoorenbeeck, Prof. dr., University Hospital, Antwerp
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: B3002021000106
Record Dates: First submitted 2023-05-09; First posted 2023-09-28 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Cystic Fibrosis
Keywords: microbiome; lactobacilli; probiotics
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Observational part of the study (No Intervention): During this part, we will collect saliva, throat and sputum samples from cystic fibrosis patients during their routine consultations in the hospital for one year.
- Probiotic group (Experimental): Daily use of a probiotic throat spray for 4 weeks
  Interventions: Biological: Probiotic throat spray

INTERVENTIONS:
Biological: Probiotic throat spray — Throat spray containing Lacticaseibacillus casei AMBR2
  Arms: Probiotic group

SUMMARY:
With this study, the investigators first want to investigate the respiratory tract microbiome of cystic fibrosis patients. To achieve this, the investigators will collect longitudinal samples of saliva, throat and sputum and process these to determine the microbial composition and compare them over a timecourse of a year. Secondly, the investigators aim to study the influence of a topical microbiome therapy (throat spray) on the microbiome of the upper and lower respiratory tract in cystic fibrosis patients after administration for 6 weeks. Bacterial and cytokine profiles of salivary, throat and sputum samples will be monitored before, during and after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis patients
* >6 years for intervention part of the study

Exclusion Criteria:

-

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Microbial composition of saliva, throat and sputum samples using 16S rRNA sequencing | Change of microbial composition over one year (observational)
Transfer of L. casei AMBR2 to the oropharyngeal cavity and lungs after administration of the throat spray | Transfer of probiotic over 6 weeks
  qPCR

SECONDARY OUTCOMES:
Changes in microbiome of the oropharyngeal region and lungs after administration of the throat spray | Baseline, 1 week, 2 weeks, 4 weeks, 6 weeks
  16S rRNA amplicon sequencing and shotgun sequencing
Influence on general health | Baseline, 1 week, 2 weeks, 4 weeks, 6 weeks
  A clinical evaluation by a specialist will be performed at the different consultations to assess general and respiratory health. A certified questionnaire including questions about the quality of life will also be filled in during each consultation.
Changes in cytokine levels (e.g. IL-10, IL-4, IL-5, IL-13) in saliva, oropharynx and sputum samples, and cytokine and antibody levels in blood samples | Baseline, 1 week, 2 weeks, 4 weeks, 6 weeks
  qPCR and/or ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Kim Van Hoorenbeeck, Principal Investigator — University Hospital, Antwerp; Sarah Lebeer, Prof., Principal Investigator — Universiteit Antwerpen
Locations (1):
- Antwerp University Hospital, Edegem, Belgium